CLINICAL TRIAL: NCT00037180
Title: Phase II, Randomized, Double-Blind, Multicenter Trial Of Celecoxib Vs Placebo For The Prevention Of Diarrhea Associated With CPT-11/5fu/LV Chemotherapy In Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: For Prevention of Diarrhea in Patients Diagnosed With Metastatic Colorectal Cancer Treated With Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IQ8-01-02-016
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Neoplasm Metastasis; Colorectal Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Celecoxib; Irinotecan; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Celecoxib
Drug: Irinotecan
Drug: 5-fluorouracil
Drug: Leucovorin

SUMMARY:
The Diarrhea Prevention with an investigational drug trial, will evaluate whether adding an investigational drug to the standard treatment for advanced colorectal cancer can reduce the amount of diarrhea a patient experiences. The standard and approved treatment for patients with metastatic colorectal cancer is repeated cycles of chemotherapy consisting of a combination of irinotecan (also known as CPT-11, Camptosar), 5-fluorouracil (also known as 5FU), and leucovorin (also known as LV). Preclinical data from animal models suggest that the investigational drug may offer an effective means for preventing CPT-11/5FU/LV-induced diarrhea. It is also hypothesized that the investigational drug-mediated anti-angiogenesis could induce a favorable tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer (either newly diagnosed or recurrent disease) with evidence of metastatic disease and present or past histological documentation of adenocarcinoma of the colon or rectum.
* Tumor must be measureable.
* Resolution of all acute toxic effects of any prior radiotherapy or surgical procedure.
* ECOG performance status 0 or 1. Age >= 18 years.
* Required baseline laboratory.
* Negative pregnancy test.
* Willingness and ability to comply with the treatment plan.

Exclusion Criteria:

* Current enrollment in another clinical trial.
* Prior adjuvant therapy for colorectal cancer <= 6 months prior to randomization.
* Prior systemic anticancer therapy or intra-arterial cytotoxic chemotherapy given as treatment for metastatic colorectal cancer.
* Known allergy to CPT-11, 5-FU, LV, celecoxib, other COX-2 inhibitors, non-steroidal anti-inflammatory drugs (NSAIDS), salicylates, or sulfonamides.
* Chronic concomitant use of full-dose aspirin, other NSAIDs or other COX-2 inhibitors for a chronic nonmalignant condition.
* A requirement for chronic concomitant use of low-dose (cardioprotective) aspirin.
* Chronic oral steroid use for treatment of a non-malignant condition.
* Known ulceration of the gastric or duodenal mucosa <= 30 days prior to randomization.
* Need for concomitant fluconazole or lithium.
* Any known significant bleeding disorder.
* Active inflammatory bowel disease or chronic diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212
Dates: Start 2002-04; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Incidence of NCI CTC grade 2-4 diarrhea during the first cycle (6 weeks) of CPT-11/5-FU/LV chemotherapy

SECONDARY OUTCOMES:
Severity of all grades of diarrhea, overall and by cycle
Duration of diarrhea, by cycle
Diarrhea grade, by day, by cycle
Stool count, by day, by cycle
Severity of asthenia (fatigue), by week.
Asthenia will be assessed with the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) scale.
Duration of asthenia, by week, as measured by the FACIT-Fatigue scale
Type, frequency, severity, timing, and relatedness of all adverse events CPT-11/5-FU/LV treatment administration as characterized by median, mean, and range of doses given; dose modifications, omissions, and delays; and actual and relative dose intensity
Compliance with celecoxib use Incidence, quantity, and duration of loperamide use
Tumor response rate (overall and confirmed)using the World Health Organization [WHO] Response Evaluation Criteria in Solid Tumors [RECIST 2000]
Serum tumor marker (carcinoembryonic antigen [CEA]) response rate (as characterized by a 50% reduction from baseline)
Time to tumor progression (TTP)
Time to treatment failure (TTF)
Survival Post-study anticancer treatment
Peak plasma levels and AUC 0-24 values for CPT-11 and its major metabolites, SN-38, SN-38 glucuronide (SN-38G), and aminopentane carboxylic acid (APC)
Inflammatory cytokines which may serve as biomarkers for cancer-related outcomes Beta-glucuronidase as a potential biomarker for tumor response
Health resource utilization (collected data to be evaluated separately from this protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Port Saint Lucie, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Saint Joseph, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=IQ8-01-02-016&StudyName=For+Prevention+of+Diarrhea+in+Patients+Diagnosed+With+Metastatic+Colorectal+Cancer+Treated+With+Chemotherapy